CLINICAL TRIAL: NCT07091071
Title: Evaluation of the CochSyn Device in Clinical Practice
Acronym: Earditech 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2025-0104
Record Dates: First submitted 2025-07-10; First posted 2025-07-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss, Sensorineural; Cochlear Hearing Loss; Cochlear Synaptopathy; DFNA9
Keywords: Auditory Evoked Potentials; Envelope Following Response; Auditory Brainstem Response; Hearing Difficulties
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Hidden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group (self-reported hearing difficulties) (Experimental): 30 subjects with self-reported hearing difficulties according to the Hearing Handicap Inventory for the Elderly - Screening Version (HHIE-s) questionnaire (score of >4)
  Interventions: Device: CochSyn device
- Control group (no self-reported hearing difficulties) (Experimental): 30 subjects without self-reported hearing difficulties according to the Hearing Handicap Inventory for the Elderly - Screening Version (HHIE-s) questionnaire (score of ≤4)
  Interventions: Device: CochSyn device
- DeaFNess Autosomal dominant 9 (DFNA9) subgroup (genetically tested and confirmed) (Experimental): 10 subjects (+3 potential drop-outs) genetically tested and confirmed to have DeaFNess Autosomal dominant 9 (DFNA9) related hearing loss
  Interventions: Device: CochSyn device

INTERVENTIONS:
Device: CochSyn device — The CochSyn device is intended for use in the evaluation of hearing-related disorders in adults using auditory evoked potentials. The CochSyn device records and analyses biopotential waveforms that can be used for hearing screening and diagnostic applications.

SUMMARY:
This study investigates a new type of auditory evoked brain potentials for the quantification and classification of peripheral hearing damage (The CochSyn Test). The study will investigate the characteristics of this new auditory evoked potential marker in a cohort of people with and without self-reported hearing difficulties and test a new type of hardware that was developed to conduct the test (the CochSyn Device) in clinical practice.

DETAILED DESCRIPTION:
Cochlear synaptopathy (CS) is a new type of sensorineural hearing loss (SNHL) and is related to ageing, noise exposure and ototoxicity. There is currently no diagnostic test of CS on the market, whereas CS is an important form of SNHL. CS occurs before the golden standard clinical hearing test (pure- tone audiogram in which participants raise their hand when hearing tones of different frequencies and the threshold of hearing is determined), shows any signs of hearing damage.

The sponsor has developed a new test, the CochSyn test that may quantify SNHL earlier than the audiogram. The newly developed test is based on auditory evoked potentials. This is a method in which an auditory stimulus is presented, and encephalogram (EEG) electrodes capture the sound-evoked brain potentials. The most popular auditory evoked potential metric to diagnose sensorineural hearing loss (SNHL) is the auditory brainstem response (ABR). Even though it can be assumed that the ABR wave-I amplitude will be sensitive to CS in humans, it may not be a differential marker for it, and hence other candidate auditory evoked potential markers for CS have been investigated. In particular, the envelope-following-response (EFR), has also been shown to be specific to CS.

The sponsor has performed several research studies on the CochSyn test that used commercially available research equipment in either humans or research animals . These data show that our marker is sensitive to ototoxic-induced CS in research animals and demonstrates an age-related decline in humans, and a superiority in terms of test-retest reliability and sensitivity compared to clinical ABR wave-I, or other evoked potential, markers. These promising data, the lack of a method to identify CS and the lack of commercially available hardware to conduct the CochSyn test in a clinical setting motivate the need for the development of the CochSyn test and device.

In this study, the sponsor wish to test the performance of its new method (the CochSyn test) in listeners with or without self-reported hearing difficulties using a newly developed hardware prototype (the CochSyn device), dedicated for the CochSyn test in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-77 years (limits included)
* Ability to fill out a questionnaire and to perform a speech intelligibility test
* Dutch or French as native language

  • Control group
* No self-reported hearing difficulties according to HHIE-s questionnaire (score of ≤4)

  • Test group
* Self-reported hearing difficulties according to HHIE-s questionnaire (score of >4)

  • Subgroup DFNA9:
* Genetically tested and confirmed to have DFNA9 related hearing loss. Note: This genetic testing was performed through standard of care testing, prior to participation in the study.

Exclusion Criteria:

* Audiometric hearing loss classifications of Moderate, Moderately severe, Severe, Profound as defined by (Clark, 1981) of the tested ear
* Asymmetrical hearing loss Note 1: Asymmetrical hearing loss is defined as an average difference of more than 15dB between both ears across the frequencies of 500, 1000, 2000 and 4000 Hz. The sum of loss in dB is divided by 4 and rounded up. A frequency not perceived is considered a loss of 120 dB.

Note 2: This exclusion criterium is not applicable for the DFNA 9 subgroup

* Tinnitus with a clinical handicap index (TFI) > 25.
* Patients with type AD, AS, B or C tympanograms
* Conductive hearing loss on the tested ear at the discretion of the investigator
* Genetic hearing loss of the tested ear Note: This exclusion criterium is not applicable for the DFNA9 subgroup.
* Congenital hearing loss of the tested ear Note: This exclusion criterium is not applicable for the DFNA9 subgroup.
* Blocked ear canal(s) of the tested ear
* Pregnant or breast-feeding
* Hearing aid user on the tested ear
* Middle ear surgery on the tested ear
* Acute ear infection of the tested ear
* Acute external auditory canal trauma on the tested ear
* Participation in session 2 of previous clinical trial NCT06114680

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Clinical performance CochSyn device: speech intelligibility | Through study completion, an average of 2,5 hours
  A significant multiple regression model that predicts speech intelligibility (quantified using the speech reception threshold) based on markers of hearing
Clinical performance CochSyn device: self-reported hearing difficulties | Through study completion, an average of 2,5 hours
  A significant multiple regression model that predicts self-reported hearing difficulties (quantified using the Hearing Handicap Inventory for the Elderly - Screening Version questionnaire) based on markers of hearing. HHIE-s score varies from 0 to 40. The higher the score the higher probability of hearing impairment.
Reliability of the CochSyn test | Through study completion, an average of 2,5 hours
  The difference between the EFR measure in a test-retest setting, where the same measurement is performed twice during the experiment.
Device related safety events of the CochSyn device | Through study completion, an average of 2,5 hours
  The cumulative rate of device related safety events throughout the study.
Technical performance of the CochSyn device | Through study completion, an average of 2,5 hours
  The cumulative rate of device deficiencies throughout the study.
Usability of the CochSyn device | Through study completion, an average of 2,5 hours
  Written feedback in form of a questionnaire and subjective comments of the test administrator on the usability of the test system for the measurements performed with the CochSyn Device after a measurement session, with regard to ease of use and comfort for both the clinician and the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Verhulst, Prof., Study Director — University Ghent
Locations (3):
- Belgium (3):
  - University Hospital Antwerp (UZA), Antwerp
  - University Hospital Ghent, Ghent
  - CHU de Liège, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van de Pol M, Verhulst S. Age-dependent traits: a new statistical model to separate within- and between-individual effects. Am Nat. 2006 May;167(5):766-73. doi: 10.1086/503331. Epub 2006 Mar 20. PMID 16671020
- [Background] Garrett M, Verhulst S. Applicability of subcortical EEG metrics of synaptopathy to older listeners with impaired audiograms. Hear Res. 2019 Sep 1;380:150-165. doi: 10.1016/j.heares.2019.07.001. Epub 2019 Jul 2. PMID 31306930
- [Background] Keshishzadeh S, Garrett M, Verhulst S. Towards Personalized Auditory Models: Predicting Individual Sensorineural Hearing-Loss Profiles From Recorded Human Auditory Physiology. Trends Hear. 2021 Jan-Dec;25:2331216520988406. doi: 10.1177/2331216520988406. PMID 33526004
- [Background] S. Verhulst, H. Van Der Biest, S. Keshishzadeh, H. Keppler, and I. Dhooge, "Supra-threshold envelope-following responses in the ageing population : an early marker of sensorineural hearing damage," in JOURNAL OF THE ACOUSTICAL SOCIETY OF AMERICA, Chicago, IL, USA, 2023, vol. 153, no. 3, Supplement, pp. A50-A50.
- [Background] N. De Poortere, W. Van Ransbeeck, S. Keshishzadeh, H. Keppler, I. Dhooge, and S. Verhulst, "Music festivals : the effect of recreational noise exposure on young adults hearing," in ARO (Association for Research in Otolaryngology) 46th Annual Midwinter Conference, Abstracts, Orlando, Florida, 2023.
- [Background] H. Van Der Biest, H. Keppler, I. Dhooge, S. Keshishzadeh, and S. Verhulst, "Cochlear synaptopathy in the ageing population," in 13th Speech in Noise Workshop, Abstracts, online, 2022.
- [Background] Verhulst S, Altoe A, Vasilkov V. Computational modeling of the human auditory periphery: Auditory-nerve responses, evoked potentials and hearing loss. Hear Res. 2018 Mar;360:55-75. doi: 10.1016/j.heares.2017.12.018. Epub 2017 Dec 28. PMID 29472062
- [Background] Vasilkov V, Caswell-Midwinter B, Zhao Y, de Gruttola V, Jung DH, Liberman MC, Maison SF. Evidence of cochlear neural degeneration in normal-hearing subjects with tinnitus. Sci Rep. 2023 Nov 30;13(1):19870. doi: 10.1038/s41598-023-46741-5. PMID 38036538